CLINICAL TRIAL: NCT01092923
Title: Nitrous Oxide and Inhalational Agent Pharmacokinetics During Anaesthetic Induction and Emergence
Brief Title: Physiological Effects of Nitrous Oxide on Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Dr Philip Peyton, Staff Anaesthetist, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03749
Record Dates: First submitted 2010-03-10; First posted 2010-03-25 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-09

CONDITIONS: Anesthesia
Keywords: Nitrous Oxide; washin; washout; second gas effect; sevoflurane; induction; emergence
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Air/Oxygen (Experimental): Sevoflurane with Air/Oxygen Mix
  Interventions: Drug: sevoflurane on air/O2
- sevoflurane in N2O/O2 (Experimental)
  Interventions: Drug: sevoflurane in N2O/O2

INTERVENTIONS:
Drug: sevoflurane on air/O2 — sevoflurane on air/O2
  Arms: Air/Oxygen
Drug: sevoflurane in N2O/O2 — sevoflurane in N2O/O2
  Arms: sevoflurane in N2O/O2

SUMMARY:
Nitrous oxide is the oldest anaesthetic agent still in routine use today. Despite huge changes in the pharmacology of volatile anaesthetic agents and intravenous anaesthetics, the unique properties of nitrous oxide have maintained its place in modern practice, where it is used in combination with other, more powerful inhaled agents, such as sevoflurane. It has useful analgesic properties, unlike the other agents used today, and its inclusion reduces the concentration of other agents required to maintain an adequate depth of anaesthesia for surgery.

In particular, its low solubility in body tissues gives it a unique pharmacokinetic profile, with rapid washin and washout from the body. It has been shown to have a similar effect on the speed of uptake of accompanying agents like sevoflurane (the "second gas effect"), which have much slower pharmacokinetics. A recent study by us suggested that this promotes faster and smoother onset of anaesthesia, as measured using the standard monitor of depth of anaesthesia (the BIS monitor). This finding requires confirmation prospectively in a larger group of patients. The investigators further hypothesise that a similar effect also exists on washout of sevoflurane at the end of the procedure, promoting quicker recovery (emergence) from anaesthesia. This has never been previously demonstrated. This information will help better define the place of nitrous oxide in achieving optimal outcomes in modern anaesthetic practice. The investigators propose to conduct a simple study to measure the effects of nitrous oxide washin and washout on exhaled concentrations of accompanying sevoflurane during both induction of anaesthesia and emergence, and identify any accompanying effect on the rate of change in depth of anaesthesia using BIS. The investigators hypothesise that the rate of fall of exhaled sevoflurane concentration at the end of anaesthesia will be more rapid in the group of patients breathing a gas mixture containing nitrous oxide, and that the rate of fall of BIS on induction and the rate of rise of BIS on emergence will be faster in the nitrous oxide group.

DETAILED DESCRIPTION:
Nitrous oxide is the oldest anaesthetic agent still in routine use today. Despite huge changes in the pharmacology of volatile anaesthetic agents and intravenous anaesthetics, the unique properties of nitrous oxide have maintained its place in modern practice, where it is used in combination with other, more powerful inhaled agents, such as sevoflurane. It has useful analgesic properties, unlike the other agents used today, and its inclusion reduces the concentration of other agents required to maintain an adequate depth of anaesthesia for surgery. In particular, its low solubility in body tissues gives it a unique pharmacokinetic profile, with rapid washin and washout from the body. It has been shown to have a similar effect on the speed of uptake of accompanying agents like sevoflurane (the "second gas effect"), which have much slower pharmacokinetics.

A recent study by us suggested that this promotes faster and smoother onset of anaesthesia, as measured using the standard monitor of depth of anaesthesia (the BIS monitor). This finding requires confirmation prospectively in a larger group of patients.

We further hypothesise that a similar effect also exists on washout of sevoflurane at the end of the procedure, promoting quicker recovery (emergence) from anaesthesia. This has never been previously demonstrated. This information will help better define the place of nitrous oxide in achieving optimal outcomes in modern anaesthetic practice.

We propose to conduct a simple study to measure the effects of nitrous oxide washin and washout on exhaled concentrations of accompanying sevoflurane during both induction of anaesthesia and emergence, and identify any accompanying effect on the rate of change in depth of anaesthesia using BIS.

Consenting adult participants will be recruited who are undergoing general anaesthesia for elective surgery anticipated to take a minimum of 1 hour and where an arterial line is considered appropriate for monitoring of blood pressure.

As, in normal practice, the decision whether to include of nitrous oxide in the anaesthetic mixture is largely discretionary on the part of the anaesthetist, and therefore allocation to either arm of the protocol is consistent with routine practice, it is intended that the patients will be approached for consent on admission to hospital for their surgery. Standard patient monitoring will be used including BIS and a 2 mL sample of blood will be taken to assess blood gas content lung function and optimise lung ventilation.

Following induction of anaesthesia, participants will receive an inhaled gas mixture containing standard concentrations of sevoflurane. They will be randomised to a treatment group where a standard concentration of nitrous oxide is included in this mixture, or a control group where nitrous oxide is not included. Monitoring and recording of exhaled gas concentrations will be made by continuous sampling of gas from the breathing circuit and computer storage. We hypothesise that the rate of fall of exhaled sevoflurane concentration at the end of anaesthesia will be more rapid in the group of patients breathing a gas mixture containing nitrous oxide, and that the rate of fall of BIS on induction and the rate of rise of BIS on emergence will be faster in the nitrous oxide group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing elective general or orthopaedic surgery under relaxant general anaesthesia anticipated to take >1 hour

Exclusion Criteria:

* Age under 18 years
* Morbid obesity BMI > 35
* Severe or moderately severe lung disease (FEV1 < 1.0L, FEV1/FVC < 50%)
* Past history of severe post-operative nausea and vomiting
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phil Peyton, MBBS, Principal Investigator — Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: December 2009 to April 2010 Location: Austin Health
Pre-assignment Details: Exclusion criteria: patients with history of severe lung disease (defined as FEV1<1.5 L or FEV1/FVC<50%), symptomatic ischemic heart disease, super obesity (BMI>45), pregnancy, prior severe post-operative nausea/vomiting, critically ill/immunocompromised, Vitamin B12/folate deficiency, or presence of any gas-filled, space-occupying lesion.
Groups:
- Sevoflurane in N2O/O2: Sevoflurane in 2:1 N2O/O2
Period: Overall Study
Arm/Group | Air/Oxygen | Sevoflurane in N2O/O2
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air/Oxygen | Sevoflurane in N2O/O2 | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 8
  >=65 years | 7 | 5 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (18) | 67 (13) | 66 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Australia | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Pa t/Pa0 Sevo (Arterial Partial Pressure of Sevoflurane), t=Time(Minutes)
Description: Rate of fall in the arterial partial pressure of sevoflurane relative to baseline at 2 minutes (Pa 2/Pa0 Sevo), 5 minutes (Pa 5/Pa0 Sevo, and 30 minutes (Pa 30/Pa0 Sevo)
Time Frame: Baseline, 2 minutes, 5 minutes, and 30 minutes after emergence
Population: based on data collected during previous pilot study investigating the magnitude of the second gas effect on sevoflurane partial pressures after anaesthesia induction, we expected an effect of roughly similar magnitude would be present during elimination of nitrous oxide.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Sevoflurane in N2O/O2: N20 with Oxygen (2:1) and Sevoflurane
- Sevoflurane in Air/O2: Air/Oxygen and Sevoflurane
Arm/Group | Sevoflurane in N2O/O2 | Sevoflurane in Air/O2
Number analyzed (Participants) | 10 | 10
ratio
  At 2 minutes | 0.32 (0.08) | 0.44 (0.13)
  At 5 minutes | 0.23 (0.07) | 0.32 (0.06)
  At 30 minutes | 0.16 (0.08) | 0.20 (0.10)

2. Secondary Outcome: Time to Eye Opening
Description: The time to eye opening to command after cessation of inhalational anaesthetic administration
Time Frame: 20 Minutes
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sevoflurane in N2O/O2 | Sevoflurane in Air/O2
Number analyzed (Participants) | 10 | 10
Minutes | 8.7 (1.3) | 11.0 (1.4)

3. Primary Outcome: PA t/PA0 Sevo (End Tidal Partial Pressure of Sevoflurane), t=Time (Minutes)
Description: Rate of fall in the end-tidal partial pressure of sevoflurane relative to baseline at 2 minutes (PA2/PA0 sevo) and 5 minutes (PA5/PA0 sevo)
Time Frame: Baseline, 2 minutes, and 5 minutes after emergence
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Sevoflurane in N2O/O2: sevoflurane with N20 and Oxygen in 2:1 mix
- Sevoflurane in Air/O2: sevoflurane in air/O2 mix
Arm/Group | Sevoflurane in N2O/O2 | Sevoflurane in Air/O2
Number analyzed (Participants) | 10 | 10
ratio
  At 2 minutes | 0.18 (0.04) | 0.22 (0.07)
  At 5 minutes | 0.14 (0.02) | 0.17 (0.06)

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Groups:
- N20 With Oxygen (2:1): sevoflurane with N20 and Oxygen in 2:1 mix
Arm/Group | N20 With Oxygen (2:1)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes